CLINICAL TRIAL: NCT00947544
Title: A Phase 2, Fixed-Sequence, Open-Label, Switch-Over Study of the Safety and Tolerability of HPN-100 Compared to Sodium Phenylbutyrate in Children 6-17 Years of Age With Urea Cycle Disorders, With a Long-Term Safety Extension
Brief Title: Study of the Safety and Tolerability of HPN-100 Compared to Sodium Phenylbutyrate in Children With Urea Cycle Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPN-100-005
Record Dates: First submitted 2009-07-24; First posted 2009-07-28 (Estimated); Results first posted 2013-12-25 (Estimated); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Urea Cycle Disorders
Keywords: Urea Cycle Disorder; UCD; GT4P; Buphenyl; hyperammonemia; sodium phenylbutyrate
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Hyperammonemia | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HPN-100 and NaPBA (Experimental): 1 week of NaPBA treatment followed by 1 week of HPN-100 treatment.
  Interventions: Drug: HPN-100; Drug: NaPBA

INTERVENTIONS:
Drug: HPN-100 — HPN-100 is a triglyceride that has a similar mechanism of action as NaPBA. It is a liquid with minimal taste and odor. Three teaspoons of HPN-100 (~17.4mL) delivers equivalent amount of PBA that 40 tablets of NapBA do.
  Other Names: GT4P, Glyceryl tri-(4-phenylbutyrate)
Drug: NaPBA — NaPBA tablets for oral administration and NaPBA powder for oral, nasogastric, or gastrostomy tube administration contain the active ingredient sodium phenylbutyrate. NaPBA is a prodrug and is rapidly metabolized to PAA, the metabolically active compound that conjugates with glutamine via acetylation to form PAGN, which is excreted by the kidneys.
  Other Names: GT4P, Glyceryl tri-(4-phenylbutyrate)

SUMMARY:
Protocol HPN-100-005 was the first study of HPN-100 in pediatric subjects with urea cycle disorders (UCDs) and was a fixed-sequence, open-label, switch over study of HPN-100 with a long-term (12 month) safety extension designed to assess the safety of HPN-100 and to prospectively assess its ability to control blood ammonia as compared with Sodium Phenylbutyrate (NaPBA). Upon DSMB review of the first ten subjects who completed the switch over part of the study, and with DSMB approval, up to an additional 20 subjects were enrolled into the safety extension part of the study. HPN-100 is a triglyceride that has a similar mechanism of action as NaPBA. It is a liquid with minimal taste and odor. Three teaspoons of HPN-100 (~17.4mL) delivers an equivalent amount of PBA to 40 tablets of NaPBA.

DETAILED DESCRIPTION:
This was a fixed-sequence, open-label, switch over study of HPN-100 with a long-term (12 month) safety extension part designed to assess the safety of HPN-100 in pediatric subjects and to prospectively assess the ability of HPN-100 to control blood ammonia compared with NaPBA.

For those subjects who participated in the switch over, NaPBA was dosed three times daily (TID) with meals during the first week and the same PBA mole-equivalent dose of HPN-100 during the second week. If there were safety concerns regarding a single-step transition from NaPBA to HPN-100, at the investigator's discretion, the transition could occur in 2 steps such that in the second week, subjects might receive 50% of the PBA equivalent dose as NaPBA and 50% as HPN-100 before receiving 100% of the PBA equivalent dose as HPN-100 in the third week. Serial blood samples were collected for PK and blood ammonia assessments after each drug reached steady state, which was achieved approximately 4 days after initiation of 100% NaPBA or HPN-100 treatment.

The subjects who completed the switch over part of the study, and up to 20 additional subjects, were offered the opportunity to continue in the study by entering the safety extension part of the study to continue receiving open-label HPN-100 for up to 12 months.

Subjects who prematurely terminated the study during the switch-over period after enrollment had safety assessments, including safety labs and a single blood sample drawn for measurement of phenylbutyrate (PBA), the active metabolite phenylacetate (PAA), and the terminal metabolite phenylacetylglutamine (PAGN). Subjects who had enrolled in the safety extension period of the study, either directly or following the switch over, but prematurely terminated the study prior to completing the extension period had Month 12 procedures performed, or at a minimum, had safety assessments including safety labs and ammonia had drawn. The time of day at which the blood sample was drawn was recorded as well as the time since the last dose of medication was taken.

Subjects followed a stable diet throughout the study, as prescribed by the investigator, and dietary compliance was recorded at each study visit for both the switch over and safety extension parts of the study.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 6-17 years old.
* Signed informed consent by subject's legally acceptable representative and assent by subject, as applicable.
* Diagnosis of urea cycle disorder (enzyme or transporter deficiency) confirmed via enzymatic, biochemical, or genetic testing.
* On a stable dose of NaPBA for a diagnosis of UCD for at least 1 week prior to the Day 1 visit.

  *Subjects who are not on a stable dose of NaPBA at the initial screening visit may be converted to a stable dose of NaPBA during the screening period and enrolled as long as they are on a stable dose of NaPBA at least 1 week prior to Day 1
* Able to perform and comply with study activities, including blood draws and urine collections.
* Negative pregnancy test for all females of childbearing potential.
* All females of childbearing age and all sexually active males must agree to use an acceptable method of contraception throughout the study.

Exclusion Criteria:

* Screening ammonia level of ≥100 μmol/L or signs and symptoms indicative of hyperammonemia; subjects may be re-screened after their ammonia is controlled, at the discretion of the investigator.
* History of 4 or more hyperammonemic events as defined in Section 3.5.1 in the preceding 12 months.
* Use of any investigational drug within 30 days of Day 1.
* Active infection (viral or bacterial) or any other condition that may increase ammonia levels.
* Any clinical or laboratory abnormality of Grade 3 or greater severity according to the CTCAE v3.0, except Grade 3 elevations in liver enzymes, defined as levels 5-20 times ULN in ALT/SGPT, aspartate aminotransferase (AST/SGOT), or gamma glutamyl transpeptidase (GGT) in a clinically stable subject.
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at increased risk by participating in this study.
* Use of any medication known to significantly affect renal clearance (e.g., probenecid) or to increase protein catabolism (e.g., corticosteroids), or other medication known to increase ammonia levels (e.g., valproate), within the 24 hours prior to Day 1 and throughout the study.
* History of QTc interval prolongation or QTc interval > 450 msec at screening or baseline.
* Known hypersensitivity to PAA or PBA.
* Liver transplant, including hepatocellular transplant.
* Currently treated with sodium benzoate or Carbaglu® (carglumic acid). At the discretion of the investigator, subjects on sodium benzoate who are otherwise eligible to participate may be switched to 100% NaPBA during the 30 day screening period as part of the study, and at least 7 days prior to Day 1 (Visit 2).
* Breastfeeding or lactating females.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (8):
- United States (7):
  - UCLA, Los Angeles, California
  - The George Washington DC Children's National Medical Center, Washington D.C., District of Columbia
  - Mount Sinai School of Medicine, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Mokhtarani M, Diaz GA, Rhead W, Berry SA, Lichter-Konecki U, Feigenbaum A, Schulze A, Longo N, Bartley J, Berquist W, Gallagher R, Smith W, McCandless SE, Harding C, Rockey DC, Vierling JM, Mantry P, Ghabril M, Brown RS Jr, Dickinson K, Moors T, Norris C, Coakley D, Milikien DA, Nagamani SC, Lemons C, Lee B, Scharschmidt BF. Elevated phenylacetic acid levels do not correlate with adverse events in patients with urea cycle disorders or hepatic encephalopathy and can be predicted based on the plasma PAA to PAGN ratio. Mol Genet Metab. 2013 Dec;110(4):446-53. doi: 10.1016/j.ymgme.2013.09.017. Epub 2013 Oct 8. PMID 24144944
- [Derived] Diaz GA, Krivitzky LS, Mokhtarani M, Rhead W, Bartley J, Feigenbaum A, Longo N, Berquist W, Berry SA, Gallagher R, Lichter-Konecki U, Bartholomew D, Harding CO, Cederbaum S, McCandless SE, Smith W, Vockley G, Bart SA, Korson MS, Kronn D, Zori R, Merritt JL 2nd, C S Nagamani S, Mauney J, Lemons C, Dickinson K, Moors TL, Coakley DF, Scharschmidt BF, Lee B. Ammonia control and neurocognitive outcome among urea cycle disorder patients treated with glycerol phenylbutyrate. Hepatology. 2013 Jun;57(6):2171-9. doi: 10.1002/hep.26058. Epub 2013 Jan 3. PMID 22961727

RESULTS

PARTICIPANT FLOW:
Groups:
- Swich Over and Safety Extension: NaPBA was dosed three times daily (TID) with during the first week and the same PBA mole-equivalent dose of HPN-100 during the second week. If there were safety concerns regarding a single-step transition from NaPBA to HPN-100, at the investigator's discretion, the transition could occur in 2 steps such that in the second week, subjects might receive 50% of the PBA equivalent dose as NaPBA and 50% as HPN-100 before receiving 100% of Serial blood samples were collected for PK and blood ammonia assessments after each drug reached steady state, which was achieved approximately 4 days after initiation of 100% NaPBA or HPN100 treatment. After the switch over, participants entered the safety extension part of the study and continued receiving open-label HPN-100 for up to 12 months.
- Safety Extension Only: Participants entered the safety extension part of the study only, and received open-label HPN-100 for up to 12 months.
Period: Switch-Over Period (2 Weeks)
Arm/Group | Swich Over and Safety Extension | Safety Extension Only
Started | 11 | 0
Completed | 11 | 0
Not Completed | 0 | 0
Period: Safety-Extension Period (12 Months)
Arm/Group | Swich Over and Safety Extension | Safety Extension Only
Started | 11 | 6 (New participants were enrolled due to DSMB approval.)
Completed | 10 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants in SO and SE: Patients who completed switch over study and enrolled safety extension study
Arm/Group | Participants in SO and SE
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10 (3.482)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 16
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Adverse Events During the Switchover Part of the Study Rate of Adverse Events (Number of Participants Showing Adverse Events)
Description: To evaluate the safety and PK characteristics of HPN-100 compared with sodium phenylbutyrate (NaPBA) in pediatric patients with urea cycle disorders (UCDs)
Time Frame: 1 week on each treatment for a total of 2 week.
Measure: Number; unit: participants
Groups:
- HPN-100: HPN-100: Patients treated with HPN-100
- NaPBA: NaPBA: Patients treated with NaPBA
Arm/Group | HPN-100 | NaPBA
Number analyzed (Participants) | 11 | 11
participants | 4 | 2

2. Secondary Outcome: Number and Causes of Hyperammonemic Events (Safety Extension)
Description: Number of Subjects with at Least One Hyperammonemic Crisis.
  Hyperammonemic crisis is defined as follows:
  • Clinical symptoms associated with ammonia of ≥ 100 µmol/L
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Pre-Enrollment (NaPBA) | Safety Extension (HPN-100)
Number analyzed (Participants) | 17 | 17
participants
  Number of subjects with at least 1 HAC | 5 | 3
  Number of Crises | 8 | 3

3. Secondary Outcome: Blood Ammonia Control
Description: To evaluate control of blood ammonia by HPN-100 compared with NaPBA in pediatric patients with UCDs.
Time Frame: Day 7 (NaPBA) and Day 14 (HPN-100)
Measure: Mean (Standard Deviation); unit: μmol∙h/L
Groups:
- HPN-100: Patients treated with HPN-100
- NaPBA: Patients treated with NaPBA
Arm/Group | HPN-100 | NaPBA
Number analyzed (Participants) | 11 | 11
μmol∙h/L | 603.83 (187.92) | 814.62 (322.36)

4. Secondary Outcome: NH3 Cmax on NaPBA vs. HPN-100 on the Last Day of Treatment With Each Drug
Description: blood samples were collected at pre-dose, 4, 8, 12, 16, 20, and 24 hour post dose on both Day 7 (NaPBA) and Day 14 (HPN-100).
Time Frame: Day 7 (NaPBA) and Day 14 (HPN-100)
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | HPN-100 | NaPBA
Number analyzed (Participants) | 11 | 11
μmol/L | 47.77 (12.8) | 55.66 (21.61)

5. Secondary Outcome: Average Ammonia Values on NaPBA vs. HPN-100 on the Last Day of Treatment With Each Drug (Switch Over)
Description: as for outcome 4
Time Frame: Day 7 (NaPBA) and Day 14 (HPN-100)
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | HPN-100 | NaPBA
Number analyzed (Participants) | 11 | 11
µmol/L | 28.68 (14.867) | 37.75 (20.310)

6. Secondary Outcome: Rate (Percentage) of Ammonia Values Above Upper Limit of Normal (ULN) on NaPBA vs. HPN-100
Description: as for outcome 4
Time Frame: Day 7 (NaPBA) and Day 14 (HPN-100)
Measure: Number; unit: percentage of sample
Units Other Than Participants: number of blood sample
Arm/Group | HPN-100 | NaPBA
Number analyzed (Participants) | 11 | 11
Number analyzed (number of blood sample) | 76 | 76
percentage of sample | 18.4 | 31.6

7. Secondary Outcome: Urinary PAGN 24-hour Excretion Values on NaPBA vs. HPN-100 (Switch Over)
Description: Urinary PAGN (phenylacetylglutamine) 24-hour excretion. Urine was collect during 0-12 hrs and 12-24 hrs.
Time Frame: Day 7 (NaPBA) and Day 14 (HPN-100)
Measure: Mean (Standard Deviation); unit: μg
Arm/Group | HPN-100 | NaPBA
Number analyzed (Participants) | 11 | 11
μg | 12501037 (56.9) | 12512426 (51.3)

8. Secondary Outcome: Plasma PAA (Phenylacetate) AUC0-24 Values on NaPBA vs. HPN-100 on on the Last Day of Treatment With Each Drug
Description: as for outcome 4
Time Frame: Day 7 (NaPBA) and Day 14 (HPN-100)
Measure: Mean (Standard Deviation); unit: μg•h/mL AUC 0-24
Arm/Group | HPN-100 | NaPBA
Number analyzed (Participants) | 11 | 11
μg•h/mL AUC 0-24 | 964 (63.6) | 773 (73.3)

9. Secondary Outcome: Plasma PBA (Phenylbutyrate) AUC0-24 Values on NaPBA vs. HPN-100 on on the Last Day of Treatment With Each Drug
Description: as for outcome 4
Time Frame: Day 7 (NaPBA) and Day 14 (HPN-100)
Measure: Mean (Standard Deviation); unit: µg*h/ml AUC 0-24
Arm/Group | HPN-100 | NaPBA
Number analyzed (Participants) | 11 | 11
µg*h/ml AUC 0-24 | 631 (44.9) | 236 (105.2)

10. Secondary Outcome: Plasma PAGN AUC0-24 Values on NaPBA vs. HPN-100 on on the Last Day of Treatment With Each Drug
Description: as for outcome 4
Time Frame: Day 7 (NaPBA) and Day 14 (HPN-100)
Measure: Mean (Standard Deviation); unit: μg*h/mL AUC 0-24
Arm/Group | HPN-100 | NaPBA
Number analyzed (Participants) | 11 | 11
μg*h/mL AUC 0-24 | 1378 (40.2) | 1015 (44.7)

11. Secondary Outcome: Quality of Life Assessed by the SF-15 Questionnaire
Description: change from baseline to Month 12.
  The SF 15 questionnaire consists of 15 questions that assess the following:
  * Physical functioning (5 questions)
  * Emotional functioning (4 questions)
  * Social functioning (3 questions)
  * School functioning (3 questions) Items were scored on a 5-point Likert scale from 0 (never) to 4 (almost always) or a 3-point scale (0 [not at all], 2 [sometimes], or 4 [a lot] for the young child self-report). Items were reverse-scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. Total score was 0-100 scale (averaged from each functional areas). In the 0-100 scale, 0 is the worst score and 100 is best score.
  Improved quality of life was shown by increased total score from baseline to Month 12.
Time Frame: 1 year
Population: Patients who completed SF-15 at baseline and Month 12 both time in the safety extension period.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: total score from SF-15 report
Groups:
- HPN-100: Patients treated with HPN-100 who completed SF-15 at baseline and Month 12
Arm/Group | HPN-100
Number analyzed (Participants) | 15
Number analyzed (total score from SF-15 report) | 30
score on a scale | 4.0 (10.67)

ADVERSE EVENTS:
Time Frame: Safety Extension period only (from Day 15 to 1 year)
Groups:
- HPN-100: HPN-100: Patient treated with HPN-100
Arm/Group | HPN-100
Serious Adverse Events (participants affected / at risk) | 3/17
Other Adverse Events (participants affected / at risk) | 4/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HPN-100 (N=17)
hyperammonemia (Metabolism and nutrition disorders) | 2
gastroenteritis (Gastrointestinal disorders) | 1
Aggression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HPN-100 (N=17)
Abdominal pain upper (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Pyrexia (General disorders) | 2
Nasopharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
ALT increased (Investigations) | 2
Anion gap increased (Investigations) | 2
AST increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperammonemia (Metabolism and nutrition disorders) | 3
Headache (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days